CLINICAL TRIAL: NCT07014592
Title: Characterization and Analysis of Evoked Cortical Responses in Participants With Medication-intractable Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Matthew S Willsey, Assistant Professor of Neurosurgery, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00258281
Record Dates: First submitted 2025-05-24; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Intractable Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Electrodes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Medication-intractable epilepsy (Experimental)
  Interventions: Device: stimulating probes and electrodes

INTERVENTIONS:
Device: stimulating probes and electrodes — Subdural electrodes and/or ball tip probes will be used intraoperatively to provide electrical stimulation to the brain.

SUMMARY:
The goal of this project is to study how the brain reacts to a small electrical signal. Researchers will be using a novel combination of recording electrodes. The researchers will measure the brain response from these electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medication intractable epilepsy who are recommended to undergo brain surgery to remove a "seizure" focus
* Can provide informed consent for the study and willing to participate

Exclusion Criteria:

* Presence of a permanent electronic implant
* Any chronic medical conditions that prevent safe placement of electrodes

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Characterization of time-frequency data | During a 20 minute research phase of a clinically indicated surgery
  From recording electrodes
Characterization of local field responses (LFPs) | During a 20 minute research phase of a clinically indicated surgery
  From recording electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Willsey, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The aspects of a plan for sharing are still under determination.